CLINICAL TRIAL: NCT01935414
Title: A Multicentre Randomised Controlled Trial Comparing the Incidence of Asymptomatic and Symptomatic Deep Vein Thrombosis Between the gekoTM Device and Thromboembolism Deterrent Stockings in Patients Recovering From Total Hip Replacement Surgery
Brief Title: Geko Neuromuscular Stimulator vs Thromboembolism Deterrent Stockings (TEDS): DVT Prevention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firstkind Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FKD-TEDS-001
Record Dates: First submitted 2013-08-28; First posted 2013-09-05 (Estimated); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- geko™ (Experimental): geko™ use continually post-surgery for 48hrs and then a minimum of 4hrs/day until discharge
  Interventions: Device: geko™ post-surgery for 48hrs then 4hrs/day until discharge.
- TEDS stockings (Active Comparator): TEDS use continually post-surgery for 48hrs and then a minimum of 4hrs/day until discharge
  Interventions: Device: TEDS post-surgery for 48hrs then 4hrs/day until discharge.

INTERVENTIONS:
Device: geko™ post-surgery for 48hrs then 4hrs/day until discharge.
  Arms: geko™
Device: TEDS post-surgery for 48hrs then 4hrs/day until discharge.
  Arms: TEDS stockings

SUMMARY:
This study hypothesises that the geko™ device is more efficient than TEDS in preventing the formation of symptomatic/asymptomatic Deep Vein Thrombosis (DVTs), post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years of age and over
2. Free of significant abnormal findings as determined by medical history (specifically an absence of DVT or haematological disorders).
3. Has not used any medications (prescribed or over-the-counter including herbal remedies) judged to be significant by the Principal Investigator during the ten (10) days preceding enrolment.
4. Able to understand the Patient Information Sheet and willing to sign the written Informed Consent Form.
5. Able and willing to follow the protocol requirements.

Exclusion Criteria:

1. Are requiring hip revision surgery
2. History or signs of previous deep or superficial vein thrombosis/pulmonary embolism.
3. Evidence of asymptomatic DVT by Duplex Ultrasound
4. Peripheral arterial disease (ABPI < 0.8), varicose veins or lower limb ulceration or ischemia.
5. Significant varicose veins, phlebitis or lower limb ulceration or ischemia. CEAP Grade 4-6. See Appendix 2
6. Recent surgery within the last 3 months (such as abdominal, gynaecological, hip or knee replacement).
7. Recent trauma to lower limb.
8. Chronic Obesity (BMI Index >40kg/m2).
9. Pregnancy.
10. Significant history of following diseases I. Cardiovascular: Recent MI (< 6 months) II. Percutaneous Coronary Intervention (PCI) with stent (< 3 months for Bare Metal Stent (BMS) and < 12 months for Drug Eluding Stent (DES) III. Moderate to severe CCF, uncontrolled AF IV. Neurological: Stroke, Hemiplegia/Paraplegia, Myopathies V. Significant dermatological conditions affecting lower limbs resulting in broken or inflamed skin particularly at the site where the device is to be fitted.

    VI. Clinically significant haematological conditions i.e. coagulation disorders, sickle cell disease VII. Psychiatric disorders
11. On LMWH/Heparin (Prophylactic/therapeutic doses) or Warfarin or warfarin stopped recently and replaced by LMWH/ Heparin
12. Long term steroid with dermatological changes
13. A pulse rate of less than 40 beats/minute
14. A sitting systolic blood pressure >180 and <100 mmHg and/or a sitting diastolic pressure of >100 mmHg.
15. Any significant illness during the four (4) weeks preceding the hip replacement surgery.
16. Participation in any clinical study during the eight (8) weeks preceding the screening period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-11-16 (Actual); Study Completion 2016-11-16 (Actual)

PRIMARY OUTCOMES:
Presence of asymptomatic DVT assessed by Duplex Ultrasound | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- BMI The Harbour Hospital, Poole, Dorset, United Kingdom

REFERENCES:
- See also: Company website — http://www.gekodevices.com/en-uk/